CLINICAL TRIAL: NCT04047446
Title: Prolonging the Interscalene Brachial Plexus Block by Adding Liposomal Bupivacaine or Preservative Free Dexamethasone to Bupivacaine: a Non-inferiority Trial
Brief Title: Liposomal Bupivacaine vs Dexamethasone ISB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-0424
Record Dates: First submitted 2019-07-03; First posted 2019-08-06 (Actual); Results first posted 2022-08-01 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Shoulder Pain
MeSH Terms: conditions — Shoulder Pain | interventions — Injections; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Liposomal bupivacaine & standard bupivacaine (Experimental)
  Interventions: Drug: Exparel 133 MG Per 10 ML Injection
- Standard bupivacaine & dexamethasone (Active Comparator)
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Exparel 133 MG Per 10 ML Injection — 10mL of 133mg liposomal bupivacaine with 5mL of 0.5% bupivacaine (15mL total)
  Other Names: Liposomal Bupivacaine
  Arms: Liposomal bupivacaine & standard bupivacaine
Drug: Dexamethasone — 15mL of 0.5% bupivacaine with 4mg of preservative-free dexamethasone will be injected
  Arms: Standard bupivacaine & dexamethasone

SUMMARY:
In this study, patients receiving shoulder arthroscopy will receive an interscalene block for pain management containing either liposomal bupivacaine and standard bupivacaine or standard bupivacaine and dexamethasone. Patients will be followed up with to determine postoperative pain and block duration.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* Age 18 years or older
* Scheduled for elective outpatient arthroscopic shoulder surgery

Exclusion Criteria:

* History of allergy to local anesthetic, or one of the study medications
* Pre-existing neurological deficits
* Psychiatric or cognitive disorders that prohibit patients from following study protocol
* History of drug or alcohol abuse
* Chronic opioid use (longer than 3 months)
* Chronic pain syndromes
* Infection at the site of injection
* Patients with severe pulmonary disease
* Herniated cervical disc, cervical myelopathy
* Contraindication for general anesthesia and/or interscalene nerve block
* Pregnancy
* Open shoulder arthrotomies.
* Non English speakers

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2019-07-11 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Kim, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures and appendices).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication
Access Criteria: Researchers who provide a methodologically sound proposal

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Liposomal Bupivacaine & Standard Bupivacaine | Standard Bupivacaine & Dexamethasone
Started | 56 | 56
Completed | 55 | 56
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liposomal Bupivacaine & Standard Bupivacaine | Standard Bupivacaine & Dexamethasone | Total
Number analyzed (Participants) | 55 | 56 | 111
Age, Continuous [Median (Inter-Quartile Range); unit: year] | 55 [48 to 61] | 49 [39 to 63] | 53 [43 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 8 | 20
  Male | 43 | 48 | 91
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 52 | 52 | 104
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 5 | 10
  White | 45 | 46 | 91
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 55 | 56 | 111
American Society of Anesthesiology Status [Count of Participants; unit: Participants] — The ASA Physical Status Classification System has been in use for over 60 years. The purpose of the system is to assess and communicate a patient's pre-anesthesia medical co-morbidities. Participants were graded by anesthesiologists pre surgery. The lower the level, the healthier the patient.
  Participants
    ASA Status I | 10 | 12 | 22
    ASA status II | 45 | 44 | 89
Body Mass Index, kg/m^2 [Mean (Standard Deviation); unit: Kg/m^2] | 27.6 (4.1) | 27.5 (4.1) | 27.6 (4.1)

OUTCOME MEASURES:

1. Primary Outcome: Numerical Rating Scale (NRS) Pain at Rest Over 72 Hours
Description: NRS pain at rest averaged over the first 72 hours. NRS pain is on a scale from 0 (no pain at all) to 10 (worst pain imaginable). Patient reported pain at 24, 48, and 72 hours are averaged to produce this number. Lower score is a better outcome.
Time Frame: First 72 hours pain
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Liposomal Bupivacaine & Standard Bupivacaine | Standard Bupivacaine & Dexamethasone
Number analyzed (Participants) | 55 | 56
score on a scale | 2.4 (1.9) | 3.4 (1.9)

2. Secondary Outcome: Numerical Rating Scale (NRS) Pain at Rest
Description: NRS pain is on a scale from 0 (no pain at all) to 10 (worst pain imaginable) and is patient reported for pain at rest. Lower score is a better outcome.
Time Frame: Postanesthesia care unit (up to 6 hours postoperative), postoperative day 1, postoperative day 2, postoperative day 3, postoperative day 4, postoperative day 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Liposomal Bupivacaine & Standard Bupivacaine | Standard Bupivacaine & Dexamethasone
Number analyzed (Participants) | 55 | 56
score on a scale
  Postanesthesia care unit (0-6 hours postoperative) | 1.3 (1.9) | 0.9 (1.8)
  Postoperative day 1 | 2.1 (2.6) | 3.0 (2.5)
  Postoperative day 2 | 2.5 (2.3) | 4.1 (2.7)
  Postoperative day 3 | 2.4 (2.2) | 3.3 (2.4)
  Postoperative day 4 | 2.5 (2.0) | 3.0 (2.2)
  Postoperative day 7 | 1.7 (2.0) | 2.3 (2.2)

3. Secondary Outcome: Numerical Rating Scale (NRS) Pain With Movement
Description: NRS pain is on a scale from 0 (no pain at all) to 10 (worst pain imaginable) and is patient reported for pain with movement. Lower score means better outcome.
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Liposomal Bupivacaine & Standard Bupivacaine | Standard Bupivacaine & Dexamethasone
Number analyzed (Participants) | 55 | 56
score on a scale
  Postanesthesia care unit (0-6 hours postoperative) | 8.9 (4.3) | 9.98 (3.2)
  Postoperative day 1 | 4.0 (3.1) | 4.3 (3.1)
  Postoperative day 2 | 4.1 (2.9) | 5.6 (3.1)
  Postoperative day 3 | 4.0 (2.7) | 5.3 (2.3)
  Postoperative day 4 | 4.0 (2.8) | 4.9 (2.4)
  Postoperative day 7 | 3.9 (2.6) | 4.7 (2.5)

4. Secondary Outcome: Opioid Consumption
Description: Opioid consumption, measured in oral morphine equivalents
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: Oral Morphine Equivalents (mg)
Arm/Group | Liposomal Bupivacaine & Standard Bupivacaine | Standard Bupivacaine & Dexamethasone
Number analyzed (Participants) | 55 | 56
Oral Morphine Equivalents (mg)
  Postanesthesia care unit (0-6 hours postoperative) | 1.8 (4.5) | 1.7 (4.6)
  Postoperative day 1 | 4.8 (8.6) | 8.1 (10.4)
  Postoperative day 2 | 12.3 (15.6) | 18.2 (20.8)
  Postoperative day 3 | 8.9 (12.5) | 13.2 (14.0)
  Postoperative day 4 | 6.9 (13.8) | 9.7 (15.5)
  Postoperative day 7 | 3.7 (7.4) | 3.3 (7.2)

5. Secondary Outcome: Patient Satisfaction With Pain Management: Scale
Description: Patient reported satisfaction on a scale of 0 (not satisfied) to 10 (complete satisfaction). This is patient opinionated and is reflective with patient contentedness with their pain management. Higher scores indicate greater satisfaction
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Liposomal Bupivacaine & Standard Bupivacaine | Standard Bupivacaine & Dexamethasone
Number analyzed (Participants) | 55 | 56
score on a scale
  Postanesthesia care unit (0-6 hours postoperative) | 9.4 (1.3) | 9.8 (0.5)
  Postoperative day 1 | 9.3 (1.4) | 9.2 (1.6)
  Postoperative day 2 | 8.9 (2.1) | 8.6 (1.8)
  Postoperative day 3 | 9.2 (1.4) | 8.6 (1.7)
  Postoperative day 4 | 9.1 (1.2) | 8.5 (1.7)
  Postoperative day 7 | 9.1 (1.5) | 8.4 (2.1)

6. Secondary Outcome: Brief Pain Inventory Short-form
Description: The Brief Pain Inventory (BPI) rapidly assesses the severity of pain and its impact on functioning. Higher scores indicate more pain. The minimum value is 0, the maximum value is 10. A lower score is a better outcome. This score is an average of the following measures on a 0-10 scale: General activity, Mood, Walking ability, Normal work, Relations to People, Sleep Quality, and Enjoyment of life.
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Liposomal Bupivacaine & Standard Bupivacaine | Standard Bupivacaine & Dexamethasone
Number analyzed (Participants) | 55 | 56
score on a scale
  Postanesthesia care unit (0-6 hours postoperative) | 1.2 (2.0) | 0.6 (1.4)
  Postoperative day 1 | 1.4 (2.0) | 1.8 (2.3)
  Postoperative day 2 | 2.4 (2.3) | 3.6 (2.5)
  Postoperative day 3 | 2.2 (2.0) | 3.4 (2.1)
  Postoperative day 4 | 2.5 (2.3) | 3.6 (2.1)
  Postoperative day 7 | 2.2 (2.1) | 2.9 (2.1)

7. Secondary Outcome: Duration of Analgesic Block
Description: Patients are contacted and asked questions regarding their motor strength and sensation in their shoulder. Patients are asked "When did your pain relief from the block completely wear off?" This indicates the block duration.
Time Frame: 24, 48, 72, 96 (if needed) hours postoperatively
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Liposomal Bupivacaine & Standard Bupivacaine | Standard Bupivacaine & Dexamethasone
Number analyzed (Participants) | 55 | 56
Hours | 26 [20 to 42] | 27 [20 to 39]

8. Secondary Outcome: Sensory Resolution
Description: Patients are contacted and asked questions regarding their motor strength and sensation in their shoulder.
Time Frame: 24, 48, 72, 96 (if needed) hours postoperatively
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Liposomal Bupivacaine & Standard Bupivacaine | Standard Bupivacaine & Dexamethasone
Number analyzed (Participants) | 55 | 56
Hours | 27 [21 to 44] | 31 [20 to 42]

9. Secondary Outcome: Motor Block Resolution
Description: Patients are contacted and asked questions regarding their motor strength and sensation in their shoulder.
Time Frame: 24, 48, 72, 96 (if needed) hours postoperatively
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Liposomal Bupivacaine & Standard Bupivacaine | Standard Bupivacaine & Dexamethasone
Number analyzed (Participants) | 55 | 56
Hours | 27 [21 to 48] | 27 [19 to 40]

10. Secondary Outcome: Time to Readiness for Discharge
Description: Time to readiness for PACU discharge was evaluated every 15min using the Post Anesthetic Discharge Scoring System.
Time Frame: Postanesthesia care unit (0-6 hours postoperative)
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Liposomal Bupivacaine & Standard Bupivacaine | Standard Bupivacaine & Dexamethasone
Number analyzed (Participants) | 55 | 56
minutes | 90 [60 to 119] | 90 [75 to 119]

11. Secondary Outcome: Postanesthesia Care Unit Length of Stay
Description: Total length of PACU stay as defined by time of PACU admission to PACU discharge.
Time Frame: Postanesthesia care unit (0-6 hours postoperative)
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Liposomal Bupivacaine & Standard Bupivacaine | Standard Bupivacaine & Dexamethasone
Number analyzed (Participants) | 55 | 56
minutes | 163.5 [138 to 197] | 163 [145 to 197]

ADVERSE EVENTS:
Time Frame: Up to 14 days following surgery
Description: At Risk patients for the Liposomal Bupivacaine group were 55 in count. However, due to lost to follow up, 43 of the 55 patients were analyzed for POD7-POD 14. At Risk patients for the Dexamethasone ISB group were 56 in count. However, due to lost to follow up, only 42 patients were able to be analyzed for POD7-POD14.
Arm/Group | Liposomal Bupivacaine & Standard Bupivacaine | Standard Bupivacaine & Dexamethasone
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/56
Other Adverse Events (participants affected / at risk) | 6/55 | 3/56
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Liposomal Bupivacaine & Standard Bupivacaine (N=55) | Standard Bupivacaine & Dexamethasone (N=56)
Postoperative neurologic symptoms at 7 days after surgery (Nervous system disorders) | 6/43 | 3/42 — Includes the presence of one or multiple: numbness, tingling, weakness, stiffness, or coldness of hand and/or finger tips, wrist, elbow, arm. Events were monitored/assessed in such a manner that the specific Adverse Event Terms cannot be separated
Postoperative neurologic symptoms at 14 days after surgery (Nervous system disorders) | 0/43 | 0/42 — Includes the presence of one or multiple: numbness, tingling, weakness, stiffness, or coldness of hand and/or finger tips, wrist, elbow, arm. Events were monitored/assessed in such a manner that the specific Adverse Event Terms cannot be separated

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-28): https://cdn.clinicaltrials.gov/large-docs/46/NCT04047446/Prot_SAP_000.pdf